CLINICAL TRIAL: NCT04118023
Title: Improving Non-Invasive Diagnosis and Grading of Cartilage Defects in the Knee - Accuracy of Ultra High Field 7-Tesla MRI as Compared With Arthroscopy
Brief Title: 7T MRI to Evaluate Cartilage Defects in the Knee
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, Principal Investigator, The Methodist Hospital Research Institute
Other Study IDs: Pro00022554
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cartilage Injury; Knee Injuries; Arthropathy of Knee; Cartilage Damage; Knee Pain Swelling
Keywords: 7T Magnetic Resonance Imaging; Clinical; Cartilaginous Lesion
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 7T MRI Group: Patient group that receives 7 Tesla Magnetic Resonance Imaging
  Interventions: Diagnostic Test: 7 Tesla Magnetic Resonance Imaging Test

INTERVENTIONS:
Diagnostic Test: 7 Tesla Magnetic Resonance Imaging Test — MAGNETOM Terra - 7T MRI Scanner by Siemens Healthineers. Each patient enrolled will undergo the study imaging test prior to planned diagnostic knee arthroscopy.

SUMMARY:
The investigators propose to prospectively evaluate the accuracy of a novel 7-Tesla (7T) knee MRI protocol for the detection and grading of cartilage lesions in the knee, which is a significant limitation of current MRI techniques.

DETAILED DESCRIPTION:
The investigators hypothesize that 7T MRI will be ~ 80% sensitive for detection of cartilaginous lesions. This will be tested in a prospective multi-reader study of 100 patients who are scheduled to have knee arthroscopy. Patients will have two MRIs of the knee: one standard of care and one experimental 7T MRI. Subjects will visit at one time point prior to scheduled knee arthroscopy, for a session time of ~1-2 hours for a single 7T MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Knee Symptomatology
* Scheduled Arthroscopic Treatment of Knee
* Adult (equal or greater than 18 years of age)

Exclusion Criteria:

* Active infections
* Less than 18 years of age
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a single surgeon in an outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Modified Whole-Organ Magnetic Resonance Imaging Score (WORMS) | baseline
  * Modified Whole-Organ Magnetic Resonance Imaging Score (WORMS) of the knee is a validated instrument utilized to grade structural abnormalities found in MRI.
  * Only the cartilage sub-score of the full WORMS will be scored in the study. Cartilage will be scored on a range from 0-6 for 6 different regional subdivisions for a minimum score of 0 and maximum score of 36. A lower score is considered a better outcome, with a score of 0 equating to normal thickness and signal of cartilage.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Miller, MD, MPH, Study Chair — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided